CLINICAL TRIAL: NCT03871192
Title: Comparison of Facet Nerve Block Versus Intra-articular Injection in the Diagnosis and Treatment of Lumbar Facet Syndrome
Brief Title: Injections in the Diagnosis and Treatment of Lumbar Facet Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Complejo Hospitalario Universitario de Granada (Other)
Responsible Party: Principal Investigator, FERNANDO RUIZ SANTIAGO, PhD, section chief musculoskeletal radiology, Complejo Hospitalario Universitario de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0607-N-18
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Facet Joint Pain; Facet Syndrome of Lumbar Spine; Facet Joints; Degeneration
Keywords: FACET JOINTS; FACET INJECTIONS; NERVE BLOCK

STUDY DESIGN:
Intervention Model Description: the patients are randomly assigned to intraarticular injection or nerve block
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the evaluator don't know if the injection was performed inside the joint or around the nerve
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- FACET JOINT UNDER CT GUIDANCE (Experimental): Injection of the facet joint under computed tomography guidance
  Interventions: Diagnostic Test: NERVE BLOCK UNDER CT GUIDANCE; Diagnostic Test: FACET JOINT UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: FACET JOINT UNDER ULTRASOUND GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER ULTRASOUND GUIDANCE
- NERVE BLOCK UNDER CT GUIDANCE (Active Comparator): Injection of the nerve under computed tomography guidance
  Interventions: Diagnostic Test: FACET JOINT UNDER CT GUIDANCE; Diagnostic Test: FACET JOINT UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: FACET JOINT UNDER ULTRASOUND GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER ULTRASOUND GUIDANCE
- FACET JOINT UNDER FLUOROSCOPY GUIDANCE (Experimental): Injection of the facet joint under fluoroscopy guidance
  Interventions: Diagnostic Test: FACET JOINT UNDER CT GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER CT GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: FACET JOINT UNDER ULTRASOUND GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER ULTRASOUND GUIDANCE
- NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE (Active Comparator): Injection of the nerve under ultrasound guidance
  Interventions: Diagnostic Test: FACET JOINT UNDER CT GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER CT GUIDANCE; Diagnostic Test: FACET JOINT UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: FACET JOINT UNDER ULTRASOUND GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER ULTRASOUND GUIDANCE
- FACET JOINT UNDER ULTRASOUND GUIDANCE (Experimental): Injection of the facet joint under ultrasound guidance
  Interventions: Diagnostic Test: FACET JOINT UNDER CT GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER CT GUIDANCE; Diagnostic Test: FACET JOINT UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER ULTRASOUND GUIDANCE
- NERVE BLOCK UNDER ULTRASOUND GUIDANCE (Active Comparator): Injection of the nerve under computed ultrasound guidance
  Interventions: Diagnostic Test: FACET JOINT UNDER CT GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER CT GUIDANCE; Diagnostic Test: FACET JOINT UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; Diagnostic Test: FACET JOINT UNDER ULTRASOUND GUIDANCE

INTERVENTIONS:
Diagnostic Test: FACET JOINT UNDER CT GUIDANCE — injection of triamcinolone in the facet joint under CT guidance
  Other Names: facet joint; ct guidance
  Arms: FACET JOINT UNDER FLUOROSCOPY GUIDANCE; FACET JOINT UNDER ULTRASOUND GUIDANCE; NERVE BLOCK UNDER CT GUIDANCE; NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; NERVE BLOCK UNDER ULTRASOUND GUIDANCE
Diagnostic Test: NERVE BLOCK UNDER CT GUIDANCE — injection of triamcinolone around the dorsal ramus under CT guidance
  Other Names: posterior ramus; ct guidance
  Arms: FACET JOINT UNDER CT GUIDANCE; FACET JOINT UNDER FLUOROSCOPY GUIDANCE; FACET JOINT UNDER ULTRASOUND GUIDANCE; NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; NERVE BLOCK UNDER ULTRASOUND GUIDANCE
Diagnostic Test: FACET JOINT UNDER FLUOROSCOPY GUIDANCE — injection of triamcinolone in the facet joint under fluoroscopy guidance
  Other Names: facet joint; fluoroscopy guidance
  Arms: FACET JOINT UNDER CT GUIDANCE; FACET JOINT UNDER ULTRASOUND GUIDANCE; NERVE BLOCK UNDER CT GUIDANCE; NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; NERVE BLOCK UNDER ULTRASOUND GUIDANCE
Diagnostic Test: NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE — injection of triamcinolone around the dorsal ramus under fluoroscopy guidance
  Other Names: posterior ramus; fluoroscopy guidance
  Arms: FACET JOINT UNDER CT GUIDANCE; FACET JOINT UNDER FLUOROSCOPY GUIDANCE; FACET JOINT UNDER ULTRASOUND GUIDANCE; NERVE BLOCK UNDER CT GUIDANCE; NERVE BLOCK UNDER ULTRASOUND GUIDANCE
Diagnostic Test: FACET JOINT UNDER ULTRASOUND GUIDANCE — injection of triamcinolone in the facet joint under ultrasound guidance
  Other Names: facet joint; ultrasound guidance
  Arms: FACET JOINT UNDER CT GUIDANCE; FACET JOINT UNDER FLUOROSCOPY GUIDANCE; NERVE BLOCK UNDER CT GUIDANCE; NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE; NERVE BLOCK UNDER ULTRASOUND GUIDANCE
Diagnostic Test: NERVE BLOCK UNDER ULTRASOUND GUIDANCE — injection of triamcinolone around the dorsal ramus under ultrasound guidance
  Other Names: dorsal ramus; ultrasound guidance
  Arms: FACET JOINT UNDER CT GUIDANCE; FACET JOINT UNDER FLUOROSCOPY GUIDANCE; FACET JOINT UNDER ULTRASOUND GUIDANCE; NERVE BLOCK UNDER CT GUIDANCE; NERVE BLOCK UNDER FLUOROSCOPY GUIDANCE

SUMMARY:
In suspected facet joints pain, it is recommended to perform nerve blocks to establish the diagnosis with positive results being and indicator of successful of most permanent treatment of facet pain by rhizolysis. Nevertheless, the usefulness of intraarticular joint injection for diagnosis and prediction of successful neurolysis have been scarcely studied. The main purpose of this trial is to compare both methods, nerve block and intra articular injection, in diagnosis and treatment of facet joints pain.

DETAILED DESCRIPTION:
Facet joint pain is considered as a nonspecific cause of spinal pain with an estimated prevalence of 12-61% of the population. At present, there are no unanimous clinical criteria to achieve and accurate diagnosis and the imaging findings do not show a direct correlation with the clinical symptoms.

Facet syndrome treatment is also controversial and, although most clinical guidelines recommend nerve block as a diagnostic test, followed by neurolysis as therapeutic technique, there are many detractors of this therapeutic sequence.

The confusion is even greater when considering the variability of specialists who perform these techniques, the variability of methods used ranging from blind injections to injections guided by ultrasound, fluoroscopy or CT, or the amount of medication injected.

The investigators have long experience in the percutaneous treatment of pain and in the use of different imaging techniques. Although the investigators objectives are multiple, the main one is to know if there are any difference in the outcome of the facet syndrome treated by intra-articular injections and the block of the medial branch of the dorsal branch of the spinal nerve.

Along with the collaboration of other specialists the investigators want to address secondary objectives such as the usefulness of ultrasound and fluoroscopy in the treatment of facet syndrome and its comparison with those performed under CT guidance that is considered as the standard technique for its greater precision.

ELIGIBILITY:
Inclusion Criteria:

1- Lumbar facet syndrome diagnosed by the referring specialist: Rehabilitation, Traumatology or Neurosurgery 2 -Mechanical low back pain that increases with rotation and flexion-extension, without radicular irradiation.

3- failure of conservative treatment (pharmacological and physical therapy). 4-Symptoms present more than 3 months

Exclusion Criteria:

1. Previous back surgery and other ablative treatments.
2. Contraindication for the use of corticosteroid or local anesthetic.
3. Uncontrolled acute or chronic medical illness.
4. Pregnancy or lactation.
5. Presence of inflammatory arthropathy or neuropathy.
6. Wounds or skin lesions in the area.
7. Diabetes mellitus.
8. Psychiatric disorders
9. Refusal to participate in the study.
10. Demonstration by imaging techniques of other causes that could justify the symptomatology.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS score) | 1 year
  score from no pain (0) to maximum pain (10)

SECONDARY OUTCOMES:
Oswestry scale | 1 year
  score from no disability(0) to maximum disability (10)

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO RUIZSANTIAGO, PhD, Principal Investigator — HOSPITAL DE NEURO-TRAUMATOLOGIA GRANADA (VIRGEN DE LAS NIEVES)
Locations (2):
- Spain (2):
  - Complejo Hospitalario Universitario Granada, Granada, SPA
  - Hospital Neuro-Traumatologia, Granada

IPD SHARING:
Plan to Share IPD: Yes
our idea is to publish the short term results and the long term results in order to influence management of this pathology. Tables and statistical analysis will be available for review and metaanalysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 to 2 years
Access Criteria: open access